CLINICAL TRIAL: NCT06640361
Title: A Single-Arm Registrational Phase III Study of Olverembatinib in the Treatment of Patients With SDH-Deficient Gastrointestinal Stromal Tumor (POLARIS-3)
Brief Title: A Study of Olverembatinib in SDH-deficient GIST.
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Ascentage Pharma Group Inc. (Industry)
Collaborators: HealthQuest Pharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HQP1351GG301
Record Dates: First submitted 2024-10-11; First posted 2024-10-15 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: GIST
Keywords: Olverembatinib; GIST
MeSH Terms: interventions — olverembatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Olverembatinib (Experimental)
  Interventions: Drug: Olverembatinib

INTERVENTIONS:
Drug: Olverembatinib — Oral administration with meal, QOD, every 28 days for a cycle.

SUMMARY:
An international multicenter, open, single-arm pivotal registration phase III study to determine the efficacy and safety of olverembatinib in patients with SDH-deficient gastrointestinal stromal tumor (GIST) who have previously been treated with one-line therapy, and to evaluate the progression-free survival and clinical benefit rate of olverembatinib in patients with SDH-deficient GIST.

DETAILED DESCRIPTION:
This study intends to enroll patients with SDH-deficient GIST who have failed at least one systemic therapy to receive olverembatinib tablets 40mg orally administered with meals once every other day and every 28 days for a dosing cycle.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically and/or cytologically confirmed GIST, immunohistochemistry with loss of SDHB expression, and failure of at least one prior systemic therapy. Defined as disease progression or intolerable as judged by the investigator.
2. Must have at least one measurable target lesion.
3. ECOG≤ 2.
4. Expected survival of at least 3 months.
5. Adequate organ function.
6. Negative serum pregnancy test result for women of childbearing potential within 7 days prior to taking the first dose of study drug.
7. Males, women of childbearing potential, as well as their partners, voluntarily take effective contraceptive measures as specified in the protocol from the time of signing the informed consent form until at least 30 days after the last dose of study drug.
8. Prior to initiation of any screening or study-specific procedures, the patient or his/her guardian is able to understand and voluntarily sign an informed consent form approved by the Ethics Committee in writing, voluntarily and able to complete the study procedures and follow-up examinations.

Exclusion Criteria:

1. Received antitumor cytotoxic chemotherapy, radiotherapy, biologic drug therapy, immunotherapy, or other investigational agents within 14 days or less than 5 times the half-life prior to the first dose.
2. Tyrosine kinase inhibitor (TKI) therapy within 7 days prior to the first dose.
3. Use of drugs that have drug interactions with the study drug within 7 days prior to the first dose.
4. Adverse events due to prior treatment have not recovered (> NCI CTCAE v5.0 Grade 1).
5. Absorption disorder syndrome or other conditions that affect the absorption of oral medications.
6. With clinically significant, uncontrolled or active cardiovascular disease or thrombotic disease.
7. Poorly controlled hypertension after hypertension medication.
8. Severe cardiovascular and cerebrovascular diseases during previous use of TKIs.
9. Uncontrolled Hyperlipidemia.
10. Major surgery, open biopsy, or major traumatic injury within 14 days prior to initiation of study drug.
11. With brain metastases.
12. Other malignancies within 2 years.
13. Uncontrolled systemic active fungal, bacterial, and/or viral infections.
14. Female patients who are pregnant or lactating, or female patients who are expecting to become pregnant within the period of this study.
15. Any symptoms or disease of the patient, in the judgment of the investigator or sponsor, that may jeopardize their safety or interfere with the safety evaluation of the investigational drug.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-11-11 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival(PFS) rate | 36 months
  Proportion of subjects who do not experience disease progression or death after the first dose of treatment as assessed by Independent Review Committee.

SECONDARY OUTCOMES:
Plasma concentrations of olverembatinib | Cycle 2 to Cycle 3 (each cycle is 28 days)
  Blood samples will be collected to measure the plasma concentration of olverembatinib.
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0. | Through study completion,an average of 2 years.
  According to CTCAE v5.0, the number and frequency of adverse events of test drug were assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Ruihua Xu, M.D., Ph.D., Study Chair — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China